CLINICAL TRIAL: NCT03604354
Title: Safety and Efficacy of Pre-emptive Tapentadol vs Pregabalin in Post Operative Pain Following Unilateral Total Knee Arthroplasty- A Randomised, Double Blind, Active Control, Clinical Trial
Brief Title: Safety and Efficacy of Pre-emptive Tapentadol vs Pregabalin in Post Operative Pain Following Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr Debasish Hota, PROFESSOR AND HEAD OF THE DEPARTMENT PHARMACOLOGY, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IEC/AIIMSBBSR/PGTH/18/12
Record Dates: First submitted 2018-07-19; First posted 2018-07-27 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis, Knee
Keywords: OA knee,pre-emptive analgesia,TKA,Opioids,gabapentinoids
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Tapentadol; Tablets; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study will be participant and investigator blinded. Allocation concealment will be done by sequentially numbered sealed drug pouches.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pregabalin (Active Comparator): Pregabalin 150mg oral tablets before one hour before undergoing unilateral total knee arthroplasty
  Interventions: Drug: Pregabalin 150mg
- Tapentadol (Experimental): tapentadol 100mg oral tablets before one hour before undergoing unilateral total knee arthroplasty
  Interventions: Drug: Tapentadol 100 MG Oral Tablet

INTERVENTIONS:
Drug: Tapentadol 100 MG Oral Tablet — This arm will receive drugs one hour before undergoing unilateral total knee arthroplasty. Interventions tapentadol 100mg oral tablets.
  Arms: Tapentadol
Drug: Pregabalin 150mg — This arm will receive drugs one hour before undergoing unilateral total knee arthroplasty. Interventions pregabalin 150mg oral tablets.
  Arms: Pregabalin

SUMMARY:
Preemptive analgesia is a treatment modality which starts even before the surgery, so that the central sensitization is prevented due to incisional injury at the time of surgery, so it covers the period of surgery and initial post-operative period preventing the development of central sensitization.

Gabapentinoid compounds are gabapentin and pregabalin which have been extensively used in seizure disorder patient. Role of gabapentinoid compounds in the management of pain, as a pre-emptive analgesia is yet to be completely evaluated in post operative pain. Opioids have always been the preferred drugs to manage post operative pain. Since opioids have major side effects of nausea vomiting associated with its treatment their use comes with management of these side effects.

Currently, diagnostic and therapeutic approaches to manage pain experienced by individuals are limited especially because there's a lack of bio-markers predictive of therapeutic outcome. In search of an objective method for pain measurement, as pain has always been subjective and it is perceived by different people differently the study will also include finding the use of COX(cyclo-oxygenase)-2 as a bio-marker of pain in post-operative patients.

Although several randomized clinical trials and met-analyses have been conducted comparing the safety and efficacy of tapentadol or pregabalin in post-operative pain, there is no head to head clinical trial conducted comparing the preemptive use of two drugs for postoperative pain following total knee arthroplasty (TKA). Hence the present study is planned.

DETAILED DESCRIPTION:
MATERIALS AND METHODS

After approval of the institutional Ethics committee board, written informed consent will be taken from all the eligible and willing patients.

A. Study design: Randomized double blind active controlled parallel group noninferiority clinical trial.

B. Randomization: A variable block randomization. The allocation ratio will be 1:1 ratio between two interventions arms i.e. tapentadol 100 mg(milligram) and pregabalin 150 mg(milligram) orally.

C. Allocation concealment: This study will be participant and investigator blinded. Allocation concealment will be done by sequentially numbered sealed drug pouches.

D. Study site: Department of Pharmacology and Orthopedics of AIIMS, Bhubaneswar.

Selection Criteria

A. Inclusion criteria

1. Patients both males and females undergoing total knee arthroplasty surgery.
2. Patients are capable of providing an informed consent.
3. Age group between 18-75 years.

B. Exclusion criteria

1. Patients with asthma, COPD(Chronic obstructive pulmonary disease) or any other respiratory disease.
2. Persistent nausea and vomiting at time of randomization
3. Epilepsy.
4. Treated with mono amine oxidase inhibitors, tricyclic antidepressants, serotonin norepinephrine re-uptake inhibitors, gabapentinoids.
5. Patient with known neurological/ neuropsychiatric disorders.
6. Drug or alcohol abuse history
7. Opioid tolerance or opioid dependence.
8. Known history of opioid allergy or pregabalin allergy.
9. Renal disease (creatinine >1.5mg/dl)
10. Liver disease (total bilirubin >1.5mg/dl)
11. Pregnancy and lactation.
12. Cardiovascular insufficiency.
13. Patient with potential serotonin syndrome.
14. Patient with history of constipation and prone to paralytic ileus.

Study procedure, tools & evaluation

1. Consent: Patients will be explained the benefit and harm of joining the study and freedom of withdrawing from the study any moment they would like to. A full voluntary written informed consent will be obtained from each patient. Study will be conducted following the principles of Helsinki after getting written permission of the institutional ethics committee. Before enrolment of first patient in this study registration for clinical trial will be done.
2. All the patients will be screened before enrollment after eliciting detailed history they will undergo complete medical and laboratory examinations.
3. A total of 90 patients of either sex will be selected randomly and will be assigned to receive 100 mg of Tapentadol or 150mg Pregabalin orally 1hr before surgery in a double-blind manner. The patient will be assessed for pain at 0,6,12, and 24hrs, post operatively by visual analogue scale score(VAS) (0-100). Pain measurements will also be done on TOTPAR scale at 0,6,12,24 hours. Total rescue analgesic consumption also will be assessed at 24hrs post operatively. All treatment emergent adverse events will be documented. The time to 1st patient request for supplemental analgesia also will be recorded.
4. A blood sample will be obtained from each of the patients twice once at 0 hrs. and again at 6hrs post operatively to evaluate concentration of COX-2 levels by ELISA with commercially available ELISA kits.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients both males and females undergoing total knee arthroplasty surgery. 2. Patients are capable of providing an informed consent. 3. Age group between 18-75 years.

Exclusion Criteria:

* 1.Patients with asthma, COPD or any other respiratory disease. 2. Persistent nausea and vomiting at time of randomization 3. Epilepsy. 4. Treated with mono amine oxidase inhibitors, tricyclic antidepressants, serotonin norepinephrine re-uptake inhibitors, gabapentinoids.

  5. Patient with known neurological/ neuropsychiatric disorders. 6. Drug or alcohol abuse history 7. Opioid tolerance or opioid dependence. 8. Known history of opioid allergy or pregabalin allergy. 9. Renal disease (creatinine >1.5mg/dl) 10. Liver disease (total bilirubin >1.5mg/dl) 11. Pregnancy and lactation. 12. Cardiovascular insufficiency. 13. Patient with potential serotonin syndrome. 14. Patient with history of constipation and prone to paralytic ileus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety of pregabalin and tapentadol by measuring the mean difference in the mean VAS score. | Evaluated over 24hrs post unilateral total knee arthroplasty
  Visual analogue scale (VAS) from 0 to 100 mm score at 0,6,12,24 hrs. post operatively in both the groups.

SECONDARY OUTCOMES:
Comparing differences in TOTPAR scale through different time points of 24 hours Comparing differences in TOTPAR (none, mild, moderate and severe) scale through different time points of 24 hours | Recorded over 24hrs post unilateral total knee arthroplasty
  Scoring on TOTPAR scale at 0,6,12,24 hrs. post operatively in both the groups
Measuring the rescue analgesic requirement in both the groups | Recorded over 24hrs post unilateral total knee arthroplasty
  Mean difference in total analgesic consumption in both the groups post operatively
Monitoring adverse events in both the groups including post-operative nausea vomiting (PONV) | Recorded over 24hrs post unilateral total knee arthroplasty
  Frequency of nausea and vomiting in both the groups.
Percentage of adverse events in a 4-point verbal scale. | Recorded over 24hrs post unilateral total knee arthroplasty
  On a scale (None, Mild, Moderate, Severe) in both the groups.
Estimation of COX-2 at 0hrs and 6hrs post operatively in both the groups by ELISA. | In two blood samples one at 0hrs and 6hrs post operatively
  Estimated in both the groups by ELISA.
Reduction of VAS and nausea/vomiting | Evaluated at the end of 6 hours and 12 hours without nausea and vomiting
  Reduction of VAS to 3 at the end of 6 hours and 12 hours without nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Debasish Hota, MD;DM, Principal Investigator — AIIMS BHUBANESWAR
Locations (1):
- All India Institute of Medical Sciences, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noah NM, Mwilu SK, Sadik OA, Fatah AA, Arcilesi RD. Immunosensors for quantifying cyclooxygenase 2 pain biomarkers. Clin Chim Acta. 2011 Jul 15;412(15-16):1391-8. doi: 10.1016/j.cca.2011.04.017. Epub 2011 Apr 17. PMID 21530501
- [Result] Brennan F, Carr DB, Cousins M. Pain management: a fundamental human right. Anesth Analg. 2007 Jul;105(1):205-21. doi: 10.1213/01.ane.0000268145.52345.55. PMID 17578977
- [Result] Kissin I. Preemptive analgesia. Anesthesiology. 2000 Oct;93(4):1138-43. doi: 10.1097/00000542-200010000-00040. No abstract available. PMID 11020772
- [Result] Garimella V, Cellini C. Postoperative pain control. Clin Colon Rectal Surg. 2013 Sep;26(3):191-6. doi: 10.1055/s-0033-1351138. PMID 24436674
- [Result] Pogatzki-Zahn EM, Segelcke D, Schug SA. Postoperative pain-from mechanisms to treatment. Pain Rep. 2017 Mar 15;2(2):e588. doi: 10.1097/PR9.0000000000000588. eCollection 2017 Mar. PMID 29392204
- [Result] Harsoor S. Emerging concepts in post-operative pain management. Indian J Anaesth. 2011 Mar;55(2):101-3. doi: 10.4103/0019-5049.79872. No abstract available. PMID 21712862
- [Result] Jain P, Jolly A, Bholla V, Adatia S, Sood J. Evaluation of efficacy of oral pregabalin in reducing postoperative pain in patients undergoing total knee arthroplasty. Indian J Orthop. 2012 Nov;46(6):646-52. doi: 10.4103/0019-5413.104196. PMID 23325966
- [Result] Dahl JB, Moiniche S. Pre-emptive analgesia. Br Med Bull. 2004 Dec 13;71:13-27. doi: 10.1093/bmb/ldh030. Print 2004. PMID 15596866
- [Result] Meacham K, Shepherd A, Mohapatra DP, Haroutounian S. Neuropathic Pain: Central vs. Peripheral Mechanisms. Curr Pain Headache Rep. 2017 Jun;21(6):28. doi: 10.1007/s11916-017-0629-5. PMID 28432601
- [Result] Rosero EB, Joshi GP. Preemptive, preventive, multimodal analgesia: what do they really mean? Plast Reconstr Surg. 2014 Oct;134(4 Suppl 2):85S-93S. doi: 10.1097/PRS.0000000000000671. PMID 25255012
- [Result] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Result] Woolf CJ, Chong MS. Preemptive analgesia--treating postoperative pain by preventing the establishment of central sensitization. Anesth Analg. 1993 Aug;77(2):362-79. doi: 10.1213/00000539-199377020-00026. No abstract available. PMID 8346839
- [Result] Silverman RB. From basic science to blockbuster drug: the discovery of Lyrica. Angew Chem Int Ed Engl. 2008;47(19):3500-4. doi: 10.1002/anie.200704280. No abstract available. PMID 18307181
- [Result] Wang YM, Xia M, Shan N, Yuan P, Wang DL, Shao JH, Ma HW, Wang LL, Zhang Y. Pregabalin can decrease acute pain and postoperative nausea and vomiting in hysterectomy: A meta-analysis. Medicine (Baltimore). 2017 Aug;96(31):e7714. doi: 10.1097/MD.0000000000007714. PMID 28767611
- [Result] Hartrick C, Van Hove I, Stegmann JU, Oh C, Upmalis D. Efficacy and tolerability of tapentadol immediate release and oxycodone HCl immediate release in patients awaiting primary joint replacement surgery for end-stage joint disease: a 10-day, phase III, randomized, double-blind, active- and placebo-controlled study. Clin Ther. 2009 Feb;31(2):260-71. doi: 10.1016/j.clinthera.2009.02.009. PMID 19302899
- [Result] Pergolizzi J, Alon E, Baron R, Bonezzi C, Dobrogowski J, Galvez R, Jensen T, Kress HG, Marcus MA, Morlion B, Perrot S, Treede RD. Tapentadol in the management of chronic low back pain: a novel approach to a complex condition? J Pain Res. 2011;4:203-10. doi: 10.2147/JPR.S19625. Epub 2011 Jul 21. PMID 21887117
- [Result] Brune K, Patrignani P. New insights into the use of currently available non-steroidal anti-inflammatory drugs. J Pain Res. 2015 Feb 20;8:105-18. doi: 10.2147/JPR.S75160. eCollection 2015. PMID 25759598